CLINICAL TRIAL: NCT07125911
Title: COMPARISON OF THE EFFECT OF COMMON ANALGESICS ON PULPAL SENSIBILITY TESTS: A CLINICAL TRIAL
Brief Title: Effect of Common Analgesia on Pulp Sensibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Kinza Iftikhar, Dr Kinza, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Dr Kinza Iftikhar
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Irreversible Pulpitis With Apical Periodontitis
MeSH Terms: interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen 400 mg (Experimental): Participants will receive a single oral dose of 400 mg ibuprofen. Cold test and electric pulp test (EPT) will be performed on a tooth with symptomatic irreversible pulpitis and on a contralateral healthy tooth before drug administration and 30 minutes after ingestion.
  Interventions: Drug: Ibuprofen 400 mg (if necessary)
- Paracetamol 500 mg (Experimental): Participants will receive a single oral dose of 500 mg paracetamol. Cold test and electric pulp test (EPT) will be performed on a tooth with symptomatic irreversible pulpitis and on a contralateral healthy tooth before drug administration and 30 minutes after ingestion.
  Interventions: Drug: Paracetamol 500 mg

INTERVENTIONS:
Drug: Ibuprofen 400 mg (if necessary) — Single oral dose of 400 mg ibuprofen administered in a blinded capsule. Prior to dosing, baseline pulpal sensibility tests (cold test with Endo-Ice and Electric Pulp Test) and pain rating (VAS) will be recorded on a contralateral healthy tooth and the target tooth with symptomatic irreversible pulpitis. The drug is given orally and tests are repeated 30 minutes after ingestion. Participants are monitored for adverse effects. Participants who cannot take NSAIDs are excluded
  Arms: Ibuprofen 400 mg
Drug: Paracetamol 500 mg — A single oral dose of 500 mg paracetamol administered in a blinded capsule. Baseline pulpal sensibility testing (cold test with Endo-Ice and Electric Pulp Test) and pain level assessment using a Visual Analogue Scale (VAS) will be performed on both the tooth with symptomatic irreversible pulpitis and a contralateral healthy tooth prior to administration. The same tests will be repeated 30 minutes after ingestion to evaluate any masking effect on test results.
  Arms: Paracetamol 500 mg

SUMMARY:
his study will investigate whether commonly used analgesics - 400 mg ibuprofen and 500 mg paracetamol - influence the accuracy of pulpal sensibility tests (cold test and electric pulp test) in patients with symptomatic irreversible pulpitis. Analgesics are often taken prior to dental visits and may mask endodontic symptoms, affecting diagnosis. Participants will be randomly assigned to receive either ibuprofen or paracetamol in a double-blind design. Test responses and pain levels will be measured before and 30 minutes after medication to assess any masking effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe pain due to SIP

Patients with prolonged pain in response to the cold test with Endo-Ice

Patients who had not used any analgesics or CNS depressant during last 6 hours

Males and females aged 18-40

Exclusion Criteria:

* patients with American Society of Anesthesiologists physical status>1

who could not take paracetamol and ibuprofen

whose teeth did not respond to the cold test

with toothache due to periapical disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Change in pulpal sensibility test results | 30 minutes after drug
  Mean change from baseline in cold test pain score (Visual Analogue Scale, 0-10) and in Electric Pulp Test (EPT) threshold value for the tooth with symptomatic irreversible pulpitis. Tests performed on the same tooth before dosing and 30 minutes after ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kinza Iftikhar, BDS, Principal Investigator — HITEC-Institute of Medical Sciences
Locations (1):
- Hitec Ims, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36657522/